CLINICAL TRIAL: NCT02984917
Title: Anterior Transversalis Fascia Approach Versus Preperitoneal Space Approach for Inguinal Hernia Repair in Residents in Northern China: a Prospective, Multi-center, Randomized, Controlled Trial
Brief Title: Anterior Transversalis Fascia Approach Versus Preperitoneal Space Approach for Inguinal Hernia Repair in Residents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Fourth Affiliated Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Hangyu Li, Chief Physician, The Fourth Affiliated Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FourthAHChinaMU_002
Record Dates: First submitted 2016-12-01; First posted 2016-12-07 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Inguinal Hernia
Keywords: anterior transversalis fascia repair; preperitoneal repair
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anterior transversalis fascia approach (Experimental): Patients with inguinal hernia will undergo inguinal hernia repair via the anterior transversalis fascia approach.
  Interventions: Procedure: Anterior transversalis fascia approach
- preperitoneal space approach (Experimental): Patients with inguinal hernia will undergo inguinal hernia repair via the preperitoneal space approach.
  Interventions: Procedure: Preperitoneal space approach

INTERVENTIONS:
Procedure: Anterior transversalis fascia approach — Patients will undergo inguinal hernia repair via the anterior transversalis fascia approach.
  Arms: anterior transversalis fascia approach
Procedure: Preperitoneal space approach — Patients will undergo inguinal hernia repair via the preperitoneal space approach.
  Arms: preperitoneal space approach

SUMMARY:
To investigate the advantages and disadvantages of the anterior transversalis fascia approach versus the preperitoneal approach for inguinal hernia repair in residents from northern China regarding common postoperative complications (including acute and chronic pain, wound infection, rates of wound infection, hematoma, seroma, and hernia recurrence) and severe postoperative complications.

DETAILED DESCRIPTION:
History and current related studies Inguinal hernia is a common surgical disease that manifests as protrusion of abdominal cavity contents through the inguinal canal because of an abdominal wall defect. It is more common in males than in females, with an overall incidence of 5-10%. Methods for surgical repair of abdominal wall defects in the inguinal region are classified as either 'tension'repairs or 'tension-free' repairs. Herniorrhaphy through repair of the posterior wall of the inguinal canal was first described by Bassini in 1887, and is regarded as a classic surgical method.

As understanding of the anatomic location and pathophysical characteristics of inguinal hernia developed, the American surgeon Lichtenstein proposed a new concept of tension-free herniorrhaphy. This technique was quickly adopted worldwide because of its advantages including minimal invasion, technical ease, effectiveness, low complication rate, low recurrence rate, and allowance of resumption of unrestricted physical activity. The most common technique is open tension-free herniorrhaphy.

Many surgical repair methods involving patches (of varying types and materials) are available for inguinal hernia repair.

Tension-free herniorrhaphy methods include anterior transversalis fascia repair, preperitoneal repair, abdominal cavity patch repair and combined repair approaches. Lichtenstein herniorrhaphy is the representative technique of anterior transversalis fascia repair. Preperitoneal repair techniques include transabdominal preperitoneal, total extraperitoneal, and Kugel repair techniques. The combined repair approaches refer to tension-free herniorrhaphy using a modified Kugel patch and the Ultrapro hernia system.

There are few reports on the effects of different inguinal hernia repair approaches on postoperative complications, particularly regarding severe postoperative complications, in patients in northern China. The incidence of severe complications after inguinal hernia repair is relatively low, but this surgery can lead to physical impairment or organ dysfunction that greatly decreases patient quality of life and places a heavy burden on the patient's family and society. At present, there is a scarcity of clinical evidence from large-sample, randomized, controlled trials investigating the effectiveness of inguinal hernia repair via the anterior transversalis fascia approach versus the preperitoneal approach.

Adverse events and serious adverse events (SAE) According to the study protocol and clinical judgment, AE/SAE occurring after herniorrhaphy will be reported to the Department of General Surgery, the Fourth Affiliated Hospital of China Medical University.

AE refer to any adverse medical events occurring after herniorrhaphy in patients or clinical subjects. SAE refer to any adverse postoperative medical events involving one or more of the following criteria:

Death, irrespective of the cause Life-threatening event Severe or permanent disability or organ dysfunction Hemorrhage Malformation, birth defect Hospitalization or extended hospital stay Re-admission to hospital Recurrence (symptomatic) of inguinal hernia

Statistical analysis Descriptive statistics will be used to analyze the data. For measurement data, the number of patients (number of missing patients), mean, median, standard deviation, first quartile, third quartile, and maximum and minimum will be described, and 95% confidence intervals will be calculated. For counted data, the frequency and relative numbers will be described, and 95% confidence intervals will be calculated. According to whether the differences between scores before and after treatments are normally distributed, the paired t-test or Wilcoxon signed rank test will be used for comparison of measurement data in the same group. The chi-squared test or Fisher's exact test will be used for analysis of counted data, and the Wilcoxon signed rank test will be used for analysis of ranked data. The last-observation-carried-forward imputation method will be used when the effects-related visit data at the last visit are missing.

Full analysis set According to the intention-to-treat principle, patients who receive at least one treatment according to study protocol and undergo at least one evaluation regarding curative effects after baseline evaluation will be included in the full analysis set.

Curative effects analysis Full analysis set analysis of curative effects will be performed. The proportions of patients with no complications, patients with common complications, and patients with severe complications within postoperative 3 weeks will be analyzed using descriptive statistics. The chi-squared test or Fisher's exact test will be used for comparison of differences between groups. If statistical differences exist between groups, the Bonferroni method will be used to adjust the α value, and pairwise comparisons will be made.

If the change in VAS pain score after treatment meets the normality and homogeneity of variance, analysis of variance will be performed. If the statistical analysis of variance results are significant, in-depth statistical analysis will be performed, and the Bonferroni method will be used for pairwise comparisons. Otherwise, the Kruskal-Wallis test will be performed. If the statistical results of the Kruskal-Wallis test are significant, in-depth statistical analysis will be performed, and the independent Wilcoxon signed rank test will be performed. The Bonferroni method will be used to adjust P values for pairwise comparisons.

Safety evaluation Safety analysis and analysis of the incidence of postoperative complications will be performed using descriptive statistics. The chi-squared test or Fisher's exact test will be performed for comparisons between groups. If significant differences exist, the Bonferroni method will be used to adjust the α value, and in-depth pairwise comparisons will be made between groups. Vital signs and laboratory outcomes will be analyzed using descriptive statistics. The paired t-test or Wilcoxon signed rank test will be used to analyze the differences between values before and after surgery. Imaging data and electrocardiograms will be analyzed using cross tabulations.

Economic analysis Cost-utility analysis will be used for economic evaluation, and sensitivity analysis of cost and utility will be performed.

Interim analysis When an adequate number of patients are enrolled and followed-up, interim analysis will be performed. When data are included for the full analysis set and recorded in the database, the first interim analysis during the management period will be performed to check whether the core data collected are suitable for preliminary significant data analysis. According to research progression, subsequent interim analysis of all data included in the database will then be designated. After acquiring approval from the Department of General Surgery and Scientific Construction Committee, the Fourth Affiliated Hospital of China Medical University, the data collected in the Department of General Surgery, the Fourth Affiliated Hospital of China Medical University are likely to be analyzed together with the data collected from the other research centers. In accordance with applicable laws and regulations, the information on the subjects in the study will be kept confidential. The data for interim analysis will be precisely described in a statistical analysis plan. The interim analysis results will be submitted to the sponsor and the project manager in the form of a statistical analysis report, and as slides by the co-sponsors.

Sample size Investigators hypothesized that anterior transversalis fascia repair can reduce the percentage of patients with postoperative pain by 15% compared with the percentage of patients with pain before surgery. Taking α = 0.05 and power = 80%, the final effective sample size of n = 300 was calculated. Assuming a patient loss rate of 20%, investigators require 360 patients. This study is planned to be performed in more than nine institutes to investigate the effectiveness of inguinal hernia repair via the anterior transversalis fascia approach versus the preperitoneal approach in patients in northern China. Investigators plan to include at least 2,000 patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary unilateral inguinal hernia
* Aged 18-80 years
* American Society of Anesthesiologists (ASA) classification I-II
* Provision of informed consent

Exclusion Criteria:

* Severe organ dysfunction or inability to tolerate surgery
* Hernia recurrence
* Giant hernia (inner size of the hernia > 4 cm)
* Scrotal hernia
* Incarcerated inguinal hernia
* Inability to complete follow-up or questionnaire because of mental disorder or other reasons
* History of preperitoneal surgery, such as radical prostatectomy

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2017-02-06 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
VAS pain score | changes of month 1, month 3, month 12, month 24 after operation
  Visual Analogue Scale(VAS) pain score is one of the most commonly used tools for assessing pain.It comprises a 10 cm line with 0 at one end, representing no pain, and 10 at the other end, representing the worst pain imaginable; the patient places a mark on the line to indicate the degree of pain that they are experiencing.

SECONDARY OUTCOMES:
Postoperative complications | changes of month 1, month 3, month 12, month 24 after operation
  Postoperative complications including wound infection, rates of hematoma, seroma, hernia recurrence, intestinal obstruction, intestinal fistula, entocele, mesenteric thrombosis, femoral vein thrombosis, ischemic orchitis, painful ejaculation, varicocele and scrotal edema.

CONTACTS AND LOCATIONS:
Overall Officials: Hangyu Li, Ph.D, Principal Investigator — The Fourth Affiliated Hospital of China Medical University
Locations (9):
- China (9):
  - General Hospital of Benxi Steel and Iron (Group) Co., LTD, Benxi, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Hospital of Dandong City, Dandong, Liaoning
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - The 202nd Hospital of PLA, Shenyang, Liaoning
  - Fengtian Hospital of Shenyang Medical College, Shenyang, Liaoning
  - General Hospital of Shenyang Military Region, Shenyang, Liaoning
  - The Fourth Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fan Q, Zhang DW, Yang DY, Li HW, Wei SB, Yang L, Yang FQ, Zhang SJ, Wu YQ, An WD, Dai ZS, Jiang HY, Wang FR, Qiao SF, Li HY. Anterior transversalis fascia approach versus preperitoneal space approach for inguinal hernia repair in residents in northern China: study protocol for a prospective, multicentre, randomised, controlled trial. BMJ Open. 2017 Aug 31;7(8):e016481. doi: 10.1136/bmjopen-2017-016481. PMID 28860228